CLINICAL TRIAL: NCT02903433
Title: Effects of Avocado Intake on the Nutritional Status of Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: San Diego State University (Other); San Ysidro Health Center (Other)
Responsible Party: Principal Investigator, Matthew Allison, Primary Investigator, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 160584
Record Dates: First submitted 2016-09-02; First posted 2016-09-16 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Cardiovascular Disease
Keywords: Avocado; Cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intake Group (Experimental): Throughout the entire study, this group will be provided with 14 avocados per week and will receive 12 bi-weekly home visits over a 6-month period during which they will receive specific brochures offering "diet tips". This group will be given specific advice on avocado consumption. Each month throughout the study, we will provide opportunities for families to visit the study kitchen at the SYHC to observe the staff preparing recipes with avocado, participate in preparing recipes, and taste recipes.
  Interventions: Other: High-intake avocados; Behavioral: Diet tips; Behavioral: Avocado consumption advice
- Low Intake Group (Active Comparator): This group will receive 3 avocados per week, as well as 12 bi-weekly home visits over a 6-month period during which they will be provided with the same educational materials (i.e., "Diet Tips") as those assigned to the "High intake" group. Participants in this group will be encouraged to improve the quality of their diets, but will not be given specific advice on avocado consumption. However, each month throughout the study, we will provide opportunities for families to visit the study kitchen at the SYHC to observe the staff preparing recipes with avocado, participate in preparing recipes, and taste recipes.
  Interventions: Other: Low-intake avocados; Behavioral: Diet tips; Behavioral: Avocado consumption advice

INTERVENTIONS:
Other: High-intake avocados — Families will receive 14 avocados on a weekly basis.
  Arms: High Intake Group
Other: Low-intake avocados — Families will receive 3 avocados on a weekly basis.
  Arms: Low Intake Group
Behavioral: Diet tips — Diet tips will come from educational materials including culturally appropriate dietary and nutritional education materials, and personalized recommendations taken from http://www.choosemyplate.gov.
Behavioral: Avocado consumption advice — Recipe book with healthy recipe suggestions that include avocado.

SUMMARY:
Avocados are an excellent source of fiber, potassium, magnesium, and poly- and mono-unsaturated fats. They can be a nutrient dense component of healthful dietary patterns and have the potential to improve the cardiovascular disease (CVD) risk profiles of families in the United States (US). The proposed research plan will focus on the contribution of avocado intake to the reduction in CVD risk of US families, by examining the effects of avocado intake on the overall nutritional status of families. Of particular interest is establishing these effects in ethnic populations such as Hispanics/Latinos. On average, Hispanic/Latinos are at increased risk for metabolic diseases that predispose to CVD. This 6-month cluster randomized trial in Hispanic/Latino Americans aims to accurately determine the impact of avocados on the overall dietary pattern of their families. Future research will extend the results of the current trial to a larger sample of ethnically diverse families in order to evaluate whether sustained changes occur in nutritional, cardiovascular and metabolic health status.

DETAILED DESCRIPTION:
Specific Aim 1: To determine how avocados are incorporated into the family's dietary pattern and impact selected measures of nutritional status:

1. To determine if avocado intake substitutes for, or adds to, other sources of calories in the family diet.
2. To determine if avocado intake helps reduce between-meal snacking of family members.
3. To determine if avocados help families meet US Dietary Guidelines for recommended intake of: poly- and monounsaturated fats; vegetables; fiber; selected nutrients (vitamins C, D and E, Folate, Calcium, Magnesium, potassium, iron); lutein and other carotenoids.

Specific aim 2: To determine if increased avocado intake affects cardio-metabolic risk factors to include lipids, glucose, insulin, and HbA1c.

ELIGIBILITY:
Inclusion Criteria:

1. Be part of a family that consists of at least 3 individuals, but no more than 8, who reside in the same home
2. Self-identify as Latino or Hispanic
3. Be older than 5 years of age

Exclusion Criteria:

1. Families with members who have clinically severe chronic diseases requiring specific diets (e.g. stage IV congestive heart failure, chronic kidney disease requiring dialysis)
2. Those allergic to avocados
3. Those with LATEX allergy
4. Families who are already high consumers of avocados (i.e. more than 1 avocado per adult and more than ½ avocado per child per day);
5. Those who are unwilling to eat avocados.
6. Family members with nursing or pregnant females or females planning to become pregnant
7. Family members under the age of 5 years will not be counted toward the number of family members who will be expected to participate in the intervention (i.e., adhere to healthy diet tips or consume avocados)
8. Families intending to move, or which include family members intending to move, within the next 6 months

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
Change in family energy consumption at 3 and 6 months | 3 months and 6 months
Change in distribution of macro and micronutrient intake at 6 months | 3 months and 6 months

SECONDARY OUTCOMES:
Change in cardio-metabolic risk factors by serum lipids at 6 months | 3 months and 6 months
Change in cardio-metabolic risk factors by insulin at 6 months | 3 months and 6 months
Change in cardio-metabolic risk factors by glucose at 6 months | 3 months and 6 months
Change in cardio-metabolic risk factors by computation of homeostasis model assessment at 6 months | 3 months and 6 months
Change in nutritional status by red blood cell fatty acid composition at 6 months | 3 months and 6 months
Change in nutritional status by red blood cell magnesium at 6 months | 3 months and 6 months
Change in nutritional status by serum total and fractionated carotenoids at 6 months | 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthew A Allison, MD, MPH, Principal Investigator — University of California, San Diego
Locations (1):
- South Bay Latino Research Center, Chula Vista, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Allen TS, Doede AL, King CMB, Pacheco LS, Talavera GA, Denenberg JO, Eastman AS, Criqui MH, Allison MA. Nutritional Avocado Intervention Improves Physical Activity Measures in Hispanic/Latino Families: A Cluster RCT. AJPM Focus. 2023 Sep 20;2(4):100145. doi: 10.1016/j.focus.2023.100145. eCollection 2023 Dec. PMID 37941823
- [Derived] VanEvery H, Pacheco LS, Sun E, Allison MA, Gao X. The impact of avocado intake on anthropometric measures among Hispanic/Latino children and adolescents: A cluster randomized controlled trial. Clin Nutr ESPEN. 2023 Aug;56:94-103. doi: 10.1016/j.clnesp.2023.04.020. Epub 2023 May 3. PMID 37344091